CLINICAL TRIAL: NCT01646814
Title: A Randomized, Blinded, Endoscopic Evaluation of Upper GI Ulceration Induced by PL2200 Versus Aspirin in At-Risk Subjects
Brief Title: Evaluation of Upper GI Ulceration Induced by PL2200 Versus Aspirin in At-Risk Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PL-ASA-005
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Gastroduodenal Ulceration
Keywords: Healthy volunteer; comparison of incidence of; treatment groups.
MeSH Terms: interventions — aspirin-phosphatidylcholine; Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PL2200 (Experimental): Investigational product, PL2200
  Interventions: Drug: PL2200
- Aspirin tablets (Active Comparator): Active comparator, 325 mg aspirin tablets
  Interventions: Drug: Aspirin tablets

INTERVENTIONS:
Drug: PL2200 — PL2200, containing 325 mg aspirin active ingredient
  Other Names: PL-ASA
  Arms: PL2200
Drug: Aspirin tablets — 325 mg aspirin tablets (USP)
  Arms: Aspirin tablets

SUMMARY:
This trial is a Phase 2, randomized, controlled study to compare the degree of mucosal injury after the oral administration of an investigational product, PL2200, and a marketed 325 mg immediate-release aspirin product.

DETAILED DESCRIPTION:
Each group will be treated with either an immediate-release aspirin tablet or PL2200 capsule at 325 mg per day for 6 weeks, and evaluated via an endoscope for any gastrointestinal injury that may have been caused by study medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, ≥50 and ≤75 years of age.
* No endoscopically observed baseline gastrointestinal lesions.

Exclusion Criteria:

* Baseline gastrointestinal lesions or abnormal screening/baseline laboratory parameters deemed clinically significant by the Investigator.
* Significant history of substance abuse or uncontrolled acute or chronic medical illness.
* Active H. pylori infection.
* Current use of low-dose aspirin for cardioprevention, or other ulcerogenic medications, gastroprotective, or anti-platelet agents.
* Hypersensitivity to aspirin or other NSAIDs.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Jupiter, Florida
  - South Miami, Florida
  - Towson, Maryland
  - New York, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PL2200 | Aspirin Tablets
Started | 121 | 126
Completed | 110 | 120
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PL2200 | Aspirin Tablets | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Customized [Number; unit: participants]
  ≥ 50 and ≤ 75 years | 121 | 126 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 82 | 153
  Male | 50 | 44 | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Gastroduodenal Ulcers
Description: Cumulative Incidence of Gastroduodenal Ulcers Greater than or equal to 3 mm in length with unequivocal depth
Time Frame: 42 Days
Population: Per protocol population (ie, Treated with ≥1 dose and Day 7 dose administered and endoscopy performed and ≥85% compliant)
Measure: Number; unit: participants
Arm/Group | PL2200 | Aspirin Tablets
Number analyzed (Participants) | 113 | 119
participants | 28 | 34

2. Secondary Outcome: Number of Subjects With Erosion and Ulcers
Description: >5 erosions or ulcers 3 mm or greater in length with unequivocal depth, by endoscopy
Time Frame: 42 days
Population: Full analysis set population, as randomized. Subjects treated with at least one dose of study drug and day 7 endoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | PL2200 | Aspirin Tablets
Number analyzed (Participants) | 119 | 121
Participants | 56 | 76
Statistical Analysis 1: Comparison: PL2200 vs Aspirin Tablets; Test type: Superiority; p = 0.019, Chi-squared

ADVERSE EVENTS:
Description: Safety Population: participants treated with ≥ 1 dose
Arm/Group | PL2200 | Aspirin Tablets
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/126
Other Adverse Events (participants affected / at risk) | 60/121 | 68/126
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL2200 (N=121) | Aspirin Tablets (N=126)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 9 (9)
Gastric Ulcer (Gastrointestinal disorders) | 26 (26) | 31 (31)
Oesophagitis (Gastrointestinal disorders) | 9 (9) | 13 (13)
Headache (Nervous system disorders) | 15 (15) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days